CLINICAL TRIAL: NCT01225965
Title: An Efficacy and Feasibility Study to Investigate the Effect of Ectoin® Inhalation Solution (EIL) in Subjects With Inflammation and Airway Obstruction Followed by a Long Term Study Extension on the Prevention of Lung Function Decline
Brief Title: Efficacy and Feasibility of Ectoin® Inhalation Solution in Inflammatory Obstruction and Ageing of the Lung
Acronym: EFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPL-015
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: COPD; Particulate Matter Induced Inflammation of the Lung
Keywords: Particulate Matter induced inflammation of the lung
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EIL05, Inhalation (Experimental)
  Interventions: Device: Ectoin Inhalation Solution
- Placebo, 0,9% NaCl (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Ectoin Inhalation Solution — Once daily inhalation of Ectoin Inhalation Solution
  Arms: EIL05, Inhalation
Device: Placebo — Once daily inhalation of Placebo Inhalation Solution
  Arms: Placebo, 0,9% NaCl

SUMMARY:
To investigate the physical inflammation inhibition effects of EIL (Ectoin-Hydro-Complex) in subjects of the established SALIA-cohort and the preventive effects on lung function decline.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females (75 - 80 years)
* FEV1/FVC < 0,77 (in the investigation 2007/2008)
* Inflammatory markers TFN-alpha > median or neutrophilic granulocytes > median (investigation 2007/2008)
* Non smokers or ex smokers who have stopped smoking for longer than 6 months

Exclusion Criteria:

* Participation in another clinical study in the previous month
* Severe concomitant disease which may have an impact on the study participation
* Hypersensitivity against Ectoin
* Myocardial infarction or apoplexy within the last year
* Uncontrolled hypertension: systolic blood pressure >200 mmHg or diastolic pressure >120 mmHg
* Known aortic aneurysm
* Other respiratory diseases (e.g. cystic fibrosis, alpha-1-Antitrypsin deficiency, sarcoidosis, allergic alveolitis, tuberculosis, etc.)
* Patients who have had treatment with live attenuated vaccinations within 14 days prior to screening visit (Inactivated influenza vaccination is acceptable, provided it is not administered within 7 days prior to screening visit)
* on investigators decision

Ages: 75 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Reduction of inflammatory markers considered to be indicative for the protective efficacy of EIL in pulmonary inflammation in COPD | Baseline and 28 days after treatment start
  Change of biomarkers in spautum, exhaled breath condensate and serum after treatment compared to baseline.

SECONDARY OUTCOMES:
Vital signs | Baseline and 28 days after treatment start
Reduction of lung function decline | Baseline and 28 days after treatment start
Change in Quality of life | Baseline and 28 days after treatment start
Need for rescue medication | 28 days (during treatment phase)
Occurence of adverse events | 28 days (during treatment phase)
Lung function parameters | 28 days (during treatment phase)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für umweltmedizinische Forschung, Düsseldorf, Germany

REFERENCES:
- See also: Website of the Institut für umweltmedizinische Forschung — http://www.iuf.uni-duesseldorf.de/englisch/home-e.htm